CLINICAL TRIAL: NCT03385629
Title: Multi-Level Interventions to Reduce Caries Disparities in Primary Care Settings
Brief Title: Providers Against Cavities in Children's Teeth
Acronym: PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Suchitra Nelson, Professor and Assistant Dean for Clinical and Translational Research, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 08-15-37; UH3DE025487-03 (NIH)
Record Dates: First submitted 2017-11-09; First posted 2017-12-28 (Actual); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Dental Caries
Keywords: Dental Care; Dental Caries; Common Sense Model of Self-Regulation
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSM theory-based Arm (Experimental): CSM theory-based didactic education and skills training Practice EMR changes
  Interventions: Behavioral: CSM theory-based didactic education and skills training; Other: Practice EMR changes
- AAP-based Arm (Active Comparator): AAP-based didactic education
  Interventions: Other: AAP-based didactic education

INTERVENTIONS:
Behavioral: CSM theory-based didactic education and skills training — Common-Sense Model of Self-Regulation (CSM) theory-based education and skills training for the provider to teach him/her to communicate core oral health facts to parents, provide a prescription to take their child to the dentist together with a list of Medicaid-accepting dentists in the area, and document the oral health encounter in EMR.
  Arms: CSM theory-based Arm
Other: AAP-based didactic education — American Academy of Pediatrics (AAP) based oral health education and follow the usual care for oral health assessment recommended by AAP guidelines.
  Arms: AAP-based Arm
Other: Practice EMR changes — Enhancements to the EMR system to include oral health documentation (four questions) which will be implemented prior to enrolling any parent/caregiver and child participants into the study.
  Arms: CSM theory-based Arm

SUMMARY:
The study is a multi-site, multi-level, and multi-component cluster randomized clinical trial (RCT) to address poor dental utilization (attendance) and untreated caries among 3-6 year old Medicaid-enrolled children attending well-child visits (WCV) in primary care settings. The focus is on addressing factors (determinants) at the socio-ecological levels of the child's environment: provider (pediatrician and nurse practitioner), practice/organization level, and parent/caregiver level. Eighteen practices will be randomized to 2 arms: A) bundled multi-level intervention consisting of: 1. training medical providers in the Common-Sense Model of Self-Regulation theory-based education so that the provider delivers to the parent/caregiver the following: i) Core oral health facts about dental caries, and ii) prescription to visit the dentist and a list of dentists accepting Medicaid; 2. Integration of oral health assessments into EMR for the provider to document in the child's medical record; versus B) Control arm of medical providers receiving the American Academy of Pediatrics (AAP) based oral health education and providing usual AAP-based care for oral health. Each arm will consist of 9 practices. Children will be followed for 24 months to determine dental utilization and changes in oral health status.

The primary aim is to examine the effectiveness of theory-based behavioral (provider-level) and implementation (practice-level) bundled interventions versus enhanced usual care (AAP based oral health education) delivered by providers at WCVs in increasing dental attendance among 3-6 year old Medicaid-enrolled children. The secondary aims are to 1) assess the effectiveness of interventions on secondary outcomes (e.g. development of new caries, changes in oral hygiene, oral health quality of life, frequency of sweet snacks and beverages, cost), 2) assess potential mediators and moderators to investigate the pathways through which the multi-level interventions affect child primary and secondary outcomes, and 3) assess the adoption, reach, fidelity, and maintenance of providers and practices that affect child primary and secondary outcomes.

The hypothesis is that theory-based behavioral (provider-level) and implementation (practice-level) bundled interventions delivered by providers at WCVs will increase dental attendance among 3-6 year old Medicaid-enrolled children versus enhanced usual care (AAP based oral health education) delivered by providers at WCVs.

DETAILED DESCRIPTION:
Study Design:

This study will utilize a cluster randomized clinical trial design (Phase III) in primary care settings. Eighteen practices will be randomized to 2 arms: A) provider-level CSM theory-based didactic and skills training to deliver oral health facts to parents, a prescription and a list of dentists accepting Medicaid + practice-level EMR changes for documenting oral health; B) AAP based didactic training with no provision of resources or changes to the practice EMR. Arm A parents/caregivers will receive oral health facts and prescription to take their child to the dentist and improve oral health behaviors in the home, while Arm B parent/caregivers will receive usual AAP-based care for oral health. Each arm will consist of 9 practices (n= 18), 33 to 34 providers (n= 67), and 512 parent/caregiver and child dyads (n= 1024). Each parent/caregiver and child dyads will be recruited at the first WCV and then followed for two consecutive WCVs (for a 24 month duration). Each provider will complete training prior to enrolling any parent/caregiver and will participate in the study for a total of 24 months duration. Immediately after randomization of practices, recruitment will be rolled-out, i.e. parent/caregivers will be recruited during a 3-month period in 6 practices at a time, with recruitment at all 18 practices expected to be completed in 9 months.

The primary outcome is receipt of dental care assessed through data abstracted from Medicaid claims files, clinical dental screenings and parent/caregiver Dental Attendance Questionnaire responses. The secondary outcomes are development of new caries, changes in oral health behaviors and oral health quality of life, dental care costs, and implementation of the interventions.

Participants:

Subjects will be pediatric providers (Pediatricians/Nurse Practitioners) and parent/caregivers and their 3-6 year old Medicaid-enrolled children from 18 primary care practices located in 6 counties in NE Ohio. The study is offered to all pediatricians/nurse practitioners in the recruited practices and will be offered to all eligible caregivers and their children excluding those with serious medical or behavioral conditions which would preclude them from participating in the dental screening. All provider and parent participants meeting the eligibility criteria will be enrolled in the study upon signing the consent form.

Procedures:

WCV #1 (Baseline): Before WCV #1, Providers (pediatrician/nurse practitioners) will receive oral health didactic education and skills training (based on study arm) to communicate core OH facts to parents/caregivers. They will complete pre- and post-tests before and after the OH didactic education session. During the well-child visit, caregivers will complete the following self-administered Baseline questionnaires: Illness Perception Questionnaire-Revised for Dental (IPQ-RD) and Parent Questionnaire. A dental hygienist will perform the child dental screening examination and study staff will record results on the ICDAS Form. During the WCV, the provider will deliver oral health facts, give a prescription to take the child to the dentist + list of local Medicaid-accepting dentists, and document oral health in EMR, based on study arm. Following the provider encounter, caregivers will provide feedback about the OH information given to them during the visit with a short self-administered Exit Questionnaire. At the end of the WCV, caregivers will be given the Follow-up IPQ-RD to be completed and returned within 2 weeks (in postage paid envelope). At six months, caregivers will report whether the child visited the dentist and also complete an annotated cost questionnaire.

WCV #2 (12 month follow-up): Before WCV #2 Providers will receive an OH didactic education booster session.

During and after the well child visit, providers and parent/child dyads will complete the same assessments and procedures done in WCV #1.

WCV #3 (24 month follow-up): There is no provider education booster session before WCV #3.

During the well child visit, providers and parent/child dyads will complete the same assessments and procedures done in WCV #1 and #2, except the IPQ-RD follow-up questionnaire. The 6 month assessments will not be completed during the third well child visit.

Analysis Plan:

Primary Statistical Analysis: For the primary outcome, the investigators will use as an overall dental attendance score the number of years (over the 24 months of follow-up) in which the child visited the dentist. This will be an ordinal outcome with possible scores of 0, 1 or 2. To assess the intervention effect, the investigators will use a generalized estimating equations (GEE) approach, with practices as clusters, based on a proportional odds marginal model. The model covariates will include an intervention indicator variable (equal to 1 for bundled intervention, 0 for enhanced usual care) and a set of baseline variables representing potential confounders. A standard error correction (for example, the method by Morel et al. 2003) will be used to adjust for a small number of clusters and 95% confidence intervals will be computed. This will be an intent-to treat analysis as all randomized participants providing the necessary measurements - regardless of any lack of compliance - will be included in the analysis.

In the event of missing data (for either year) for dental attendance, the investigators will conduct sensitivity analyses by imputing responses under conservative assumptions (favoring the null hypothesis) and re-running the analysis described above on the completed data.

Analysis of Secondary Outcomes: Summary statistics (including means and standard errors) for secondary outcomes will be calculated by intervention group. The same approach as above will be used for binary or ordinal secondary outcomes (oral hygiene, frequency of sweet snacks and beverages). Namely, ordinal outcomes for each variable will be defined that summarize outcomes over time. For continuous outcomes (e.g., OH quality of life, cost), the above method will be modified by using a linear model (identify link) for GEE, modeling the mean response over time as a summary measure. These outcomes will each be tested for normality using the Shapiro-Wilk statistic; outcomes for which normality is violated will be transformed where appropriate or an alternative model used. For count outcomes (e.g., dft accumulated over time), the investigators will use a loglinear model (log link) assuming a negative binomial or other appropriate (e.g., zero-inflated negative binomial) distribution. For proportion outcomes (e.g., dt/dft), the investigators will use GEE with a logit link, assuming the proportion follows a beta binomial or zero-inflated beta binomial distribution. Similarly, the investigators will fit appropriate GEE models to test for the effect of each implementation strategy on the corresponding outcome (e.g., % prescriptions given as a measure of adoption). As in the dental attendance analysis, the intervention indicator as well as pertinent baseline variables will be included in the model. In addition, interaction terms (baseline variables by intervention) will be included to test for possible effect modification.

For secondary analyses, a GLIMMIX model approach will be considered as an alternative, which may more easily allow for more than one cluster level if needed. Another alternative approach is to model the repeated measurements (again using GEE or GLIMMIX) which will add an additional cluster level - namely, for individuals). Goodness of fit of alternative models will be compared using QIC for GEE (or AIC for GLIMMIX).

Missing Data: In the likely event of missing responses, the investigators will first assess (In the context of repeated measures analyses) whether the data are missing completely at random (MCAR), that is, whether missingness of the given outcome is dependent only on participant baseline characteristics and not further on the observed outcome at an earlier time. This will be done by modeling missing data indicators for the repeated measurements of each outcome using a GEE (or GLIMMIX) approach with a logit link and including appropriate baseline (control) variables and the outcome at the previous time if available. The MCAR null hypothesis will be rejected if the previous outcome has a statistically significant effect on the probability of missing. A nonsignificant effect would support the use of GEE (which assumes MCAR). In addition to assessing the overall effects of the interventions, the investigators will investigate the mechanisms (or paths) through which interventions impact dental attendance.

Data Management:

The study staff will collaborate and interact with the NIH-appointed Coordinating Center (CC) to perform data management and quality control activities. Study data will be collected and stored using the REDCap platform hosted by University of California-San Francisco, the home institution of the CC. REDCap is a secure, web-based application designed to support remote data capture for research studies.

Study forms will be completed by participants on paper, and subsequently entered into REDCap by study staff, or on a tablet directly into REDCap. Paper forms will be securely stored in a locked file cabinet. Recorded audio will be deleted from the digital recording device immediately after being stored on a secure CWRU School of Dental Medicine network drive.

Data for this study will include: (1) dental screening data, (2) study questionnaires, (3) abstracted medical data, (4) abstracted Medicaid dental claims data, (5) cost data (6) data from observation/audiotaping of providers, and (7) EMR audit data. Additionally, audio recordings will be used for fidelity monitoring. Form revisions should be minimal; however, should they occur, changes will be submitted to the CC for updating and dissemination to study staff.

Quality control is primarily conducted at the study team level through internal processes of data review/data monitoring using periodic custom reports generated by the CC. The CC will assist with the design of project-specific custom reports. The CC will run regular validation reports to detect data anomalies and will work with the local project staff to resolve any data anomalies that arise during data entry. REDCap's native data resolution workflow will be used to document and fix any data anomalies. The Data Manager will also respond to data queries generated by the PI, Study Coordinator, or other study staff.

The CC will generate regular reports showing enrollment and potential data anomalies, which will be sent to PIs, Project Coordinators, and other relevant study staff.

ELIGIBILITY:
Inclusion Criteria:

Practices:

* Use Electronic Medical Record (EMR)
* Have ≥ 20% of pediatric patients covered by Medicaid

Providers:

* Pediatrician or Nurse Practitioner with a minimum of 2 patient-care days per week
* Provide signed and dated consent form

Parents or caregivers:

* Legal guardianship of Medicaid-enrolled children aged 3-6 years attending well-child visit (WCV)
* Must be ≥ 18 years
* Speak English or Spanish
* Provide signed and dated consent form
* Planning to stay in the immediate area (both parent/caregiver and child) for at least two years

Child:

* Ages 3-6 years
* Enrolled in Medicaid

Exclusion Criteria:

Child:

● Presence of any serious medical or behavioral condition (e.g. cerebral palsy, autism) that precludes participation in the dental screening

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2108 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra Nelson, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nelson S, Albert JM, Selvaraj D, Curtan S, Momotaz H, Bales G, Ronis S, Koroukian S, Rose J. Multilevel Interventions and Dental Attendance in Pediatric Primary Care: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2024 Jul 1;7(7):e2418217. doi: 10.1001/jamanetworkopen.2024.18217. PMID 38980678
- [Derived] Nelson S, Slusar MB, Curtan S, Selvaraj D, Hertz A. Formative and Pilot Study for an Effectiveness-Implementation Hybrid Cluster Randomized Trial to Incorporate Oral Health Activities into Pediatric Well-Child Visits. Dent J (Basel). 2020 Sep 1;8(3):101. doi: 10.3390/dj8030101. PMID 32882958

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included 18 primary care practices in northeast Ohio randomized into 1 of 2 arms using a restricted randomization scheme with 9 practices assigned to each arm. Providers and parent-child dyads were participants assigned to groups based on affiliated practice. 63 Providers and 1024 parent-child dyads were recruited between 11/2017 and 8/2019. 1 provider, 1 parent-child dyad were late exclusions, leaving 2108 individuals enrolled (62 providers, 1023 parent/caregivers & 1023 children).
Units Other Than Participants: Practices
Groups:
- CSM Theory-based Arm: 1. CSM theory-based didactic education and skills training for providers
     CSM theory-based didactic education and practical skills training: Common-Sense Model of Self-Regulation (CSM) theory-based education and skills training for the provider to teach him/her to communicate core oral health facts to parents, provide a prescription to take their child to the dentist together with a list of Medicaid-accepting dentists in the area, and how to document the oral health encounter in EMR.
  2. Practice EMR changes w/oral health questions
  Practice EMR changes: Enhancements to the EMR system to include oral health documentation (four questions) which will be implemented prior to enrolling any parent/caregiver and child participants into the study.
- AAP-based Arm: AAP-based didactic education (without theory-based training, skills training or EMR changes)
  AAP-based didactic education: American Academy of Pediatrics (AAP) based oral health education and follow the usual care for oral health assessment recommended by AAP guidelines.
Period: Baseline Well Child Visit 1
Arm/Group | CSM Theory-based Arm | AAP-based Arm
Started | 1061; 9 Practices (27 Providers, 517 Parent/Caregiver-child dyads (517 Parents/Caregivers, 517 children)) | 1047; 9 Practices (35 Providers, 506 Parent/Caregiver-Child Dyads (506 Parents/Caregivers, 506 Children))
Completed | 1061; 9 Practices (27 Providers, 517 Parent/Caregiver-child dyads (517 Parents/Caregivers, 517 children)) | 1047; 9 Practices (35 Providers, 506 Parent/Caregiver-Child Dyads (506 Parents/Caregivers, 506 Children))
Not Completed | 0; 0 Practices | 0; 0 Practices
Period: Follow-up Well Child Visit 2
Arm/Group | CSM Theory-based Arm | AAP-based Arm
Started | 1035; 9 Practices (27 Providers, 504 Parent/Caregiver-child dyads (504 Parents/Caregivers, 504 children) The number starting Follow-up Well Child Visit 2 is lower than the number completing Baseline Well Child Visit 1 because 13 Parents/Caregivers and 13 Children withdrew between the Well Child Visits.) | 1023; 9 Practices (35 Providers, 494 Parent/Caregiver-Child Dyads (494 Parents/Caregivers, 494 Children).The number starting this period (Well Child Visit 2) is lower than the number completing Baseline Well Child Visit 1 because 12 Parents/Caregivers and 12 Children withdrew between the Well Child Visits.)
Completed (Follow-up Well Child Visit 2) | 815; 9 Practices (21 Providers, 397 Parent/Caregiver-child dyads (397 Parents/Caregivers, 397 children)) | 860; 9 Practices (32 Providers, 414 Parent/Caregiver-Child Dyads (414 Parents/Caregivers, 414 Children).)
Not Completed | 220; 0 Practices | 163; 0 Practices
Not completed — Lost to Follow-up | 214 | 160
Not completed — Withdrawal by Subject | 6 | 3
Period: Follow-up Well Child Visit 3
Arm/Group | CSM Theory-based Arm | AAP-based Arm
Started | 1019; 9 Practices (21 Providers, 499 Parent/Caregiver-child dyads (499 Parents/Caregivers, 499 children). Participants did not have to complete WCV 2 to be eligible to complete WCV 3, therefore the number of participants starting (eligible) is higher than the number completing WCV 2. Only those who withdrew themselves prior to WCV 2 and 3 (6 providers + 18 parents/caregivers + 18 children = 42 individuals) are not included in the number started (eligible). Those lost to follow-up were not considered as withdrawn.) | 1006; 9 Practices (32 Providers, 487 Parent/Caregiver-Child Dyads (487 Parents/Caregivers, 487 Children). Participants did not have to complete WCV 2 to be eligible to complete WCV 3, therefore the number of participants starting (eligible) is higher than the number completing WCV 2. Only those who withdrew themselves prior to WCV 2 and 3 (3 Providers + 19 parents/caregivers + 19 children = 41 individuals) are not included in the number started (eligible). Those lost to follow-up were not considered as withdrawn.)
Completed | 753; 9 Practices (21 Providers, 366 Parent/Caregiver-child dyads (366 Parents/Caregivers, 366 children).) | 820; 9 Practices (32 Providers, 394 Parent/Caregiver-Child Dyads (394 Parents/Caregivers, 394 Children).)
Not Completed | 266; 0 Practices | 186; 0 Practices
Not completed — Lost to Follow-up | 266 | 186

BASELINE CHARACTERISTICS:
Population: The baseline analysis population is 2108 (62 providers, 1023 parent/caregivers and 1023 children). One provider and one parent/child dyad were late exclusions due to not meeting the inclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | CSM Theory-based Arm | AAP-based Arm | Total
Number analyzed (Participants) | 1061 | 1047 | 2108
Age, Continuous [Mean (Standard Deviation); unit: children, providers, parents: yrs] — Population: Analysis was completed separately for each group: Parents/Caregivers (1023), Children (1023), and Providers (62)
  children, providers, parents: yrs
    Children: number analyzed (Participants) | 517 | 506 | 1023
    Children | 4.70 (1.20) | 4.65 (1.11) | 4.68 (1.17)
    Parents/caregivers: number analyzed (Participants) | 517 | 506 | 1023
    Parents/caregivers | 31.73 (7.89) | 31.10 (7.02) | 31.42 (7.48)
    Providers: number analyzed (Participants) | 27 | 35 | 62
    Providers | 43.70 (10.13) | 49.43 (11.74) | 46.94 (11.35)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Analysis was completed separately for each group: Parents/Caregivers (1023), Children (1023), and Providers (62). The number analyzed differs from the overall number due to some missing data
  Participants
    Children: number analyzed (Participants) | 516 | 505 | 1021
    Children: Female | 228 | 238 | 466
    Children: Male | 288 | 267 | 555
    Parents/caregivers: number analyzed (Participants) | 515 | 506 | 1021
    Parents/caregivers: Female | 463 | 457 | 920
    Parents/caregivers: Male | 52 | 49 | 101
    Providers: number analyzed (Participants) | 27 | 35 | 62
    Providers: Female | 22 | 25 | 47
    Providers: Male | 5 | 10 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Analysis was completed separately for each group: Parents/Caregivers (1023), Children (1023), and Providers (62)
  Participants
    Children: number analyzed (Participants) | 517 | 506 | 1023
    Children: Hispanic or Latino | 28 | 48 | 76
    Children: Not Hispanic or Latino | 457 | 425 | 882
    Children: Unknown or Not Reported | 32 | 33 | 65
    Parents/caregivers: number analyzed (Participants) | 517 | 506 | 1023
    Parents/caregivers: Hispanic or Latino | 20 | 31 | 51
    Parents/caregivers: Not Hispanic or Latino | 466 | 447 | 913
    Parents/caregivers: Unknown or Not Reported | 31 | 28 | 59
    Providers: number analyzed (Participants) | 27 | 35 | 62
    Providers: Hispanic or Latino | 0 | 0 | 0
    Providers: Not Hispanic or Latino | 23 | 25 | 48
    Providers: Unknown or Not Reported | 4 | 10 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Analysis was completed separately for each group: Parents/Caregivers (1023), Children (1023), and Providers (62)
  Participants
    Children: number analyzed (Participants) | 517 | 506 | 1023
    Children: American Indian or Alaska Native | 2 | 0 | 2
    Children: Asian | 0 | 4 | 4
    Children: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Children: Black or African American | 226 | 225 | 451
    Children: White | 232 | 209 | 441
    Children: More than one race | 41 | 49 | 90
    Children: Unknown or Not Reported | 15 | 19 | 34
    Parents/caregivers: number analyzed (Participants) | 517 | 506 | 1023
    Parents/caregivers: American Indian or Alaska Native | 2 | 0 | 2
    Parents/caregivers: Asian | 1 | 3 | 4
    Parents/caregivers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Parents/caregivers: Black or African American | 223 | 215 | 438
    Parents/caregivers: White | 256 | 241 | 497
    Parents/caregivers: More than one race | 17 | 28 | 45
    Parents/caregivers: Unknown or Not Reported | 18 | 19 | 37
    Providers: number analyzed (Participants) | 27 | 35 | 62
    Providers: American Indian or Alaska Native | 0 | 0 | 0
    Providers: Asian | 2 | 3 | 5
    Providers: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Providers: Black or African American | 2 | 2 | 4
    Providers: White | 22 | 26 | 48
    Providers: More than one race | 0 | 3 | 3
    Providers: Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1061 | 1047 | 2108
dft [Mean (Standard Deviation); unit: decayed and filled teeth] — Number of decayed and filled teeth Population: Analysis population is children examined. Two children could not be examined due to behavioral issues.
  decayed and filled teeth
    number analyzed (Participants) | 516 | 505 | 1021
    (all) | 1.44 (2.45) | 1.27 (2.33) | 1.36 (2.39)
Frequency of tooth brushing [Mean (Standard Deviation); unit: number of times per day child brushes] — How often child's teeth are brushed Population: Mean number of times/day children brush. The number analyzed differs from the overall number due to some missing data
  number of times per day child brushes
    number analyzed (Participants) | 510 | 501 | 1011
    (all) | 1.87 (0.60) | 1.77 (0.62) | 1.82 (0.61)
Frequency of intake of sweet drinks [Mean (Standard Deviation); unit: Number of sugar-sweetened beverages/day] — number of sugar sweetened beverages/day Population: The number analyzed differs from overall number due to some missing data.
  Number of sugar-sweetened beverages/day
    number analyzed (Participants) | 508 | 498 | 1006
    (all) | 0.44 (0.78) | 0.51 (0.78) | 0.47 (0.78)
The Early Childhood Oral Health Impact Scale (ECOHIS) [Mean (Standard Deviation); unit: scores on a scale] — The mean overall numeric score for the ECOHIS questionnaire at baseline. This 13 item questionnaire was scored on a Likert scale ranging from 0 to 4. An overall score was calculated for each child and a mean calculated at baseline. Lower scores indicating a better oral health quality of life. Population: The number analyzed differs from the overall number due to some missing data
  scores on a scale
    number analyzed (Participants) | 507 | 502 | 1009
    (all) | 1.42 (2.91) | 1.45 (2.90) | 1.43 (2.90)

OUTCOME MEASURES:

1. Primary Outcome: Dental Attendance
Description: Receipt of any dental care (preventive and/or restorative) at approximately 24 months from baseline to the exit visit. Any dental care was defined as yes or no visit.
Time Frame: Data will be abstracted from Clinical Exams and Medicaid Claims data at baseline and the exit visit at the 24 month follow-up visit.
Population: Any child dental visits through WCV3. The number of children with Medicaid claims data was 865. The number of children with clinical examinations was 675.
Measure: Count of Participants; unit: Participants
Arm/Group | CSM Theory-based Arm | AAP-based Arm
Number analyzed (Participants) | 448 | 417
Participants
  Medicaid Claims Data | 330 | 332
  Clinical Examination Data: number analyzed (Participants) | 327 | 348
  Clinical Examination Data | 170 | 150

2. Secondary Outcome: Change in Primary Decayed and Filled Teeth
Description: dft: number of decayed, missing and filled teeth (dft) at WCV#3 minus the number at WCV#1.
Time Frame: Dental exams will assess change in dft between baseline well-child visit (WCV#1) and 24 month follow-up exit visit (well-child visit: WCV#3)
Population: The number analyzed is lower than the number enrolled at WCV1 (baseline) due to not all children having an exam at WCV3
Measure: Mean (Standard Deviation); unit: teeth
Arm/Group | CSM Theory-based Arm | AAP-based Arm
Number analyzed (Participants) | 301 | 331
teeth | 1.14 (2.45) | 1.16 (2.34)

3. Secondary Outcome: Change in Oral Hygiene-brushing
Description: Change in mean number of times per day a child in the study brushed.
Time Frame: Assessed as change between baseline well-child visit (WCV #1) and 24 month follow-up exit visit (well-child visit: WCV#3)
Population: The number analyzed is lower than the number enrolled at WCV1 (baseline) due to some missing data or the study visit not being completed for WCV3
Measure: Mean (Standard Deviation); unit: mean number of times/day child brushes
Arm/Group | CSM Theory-based Arm | AAP-based Arm
Number analyzed (Participants) | 359 | 375
mean number of times/day child brushes | -0.01 (0.63) | -0.04 (0.62)

4. Secondary Outcome: Change in Diet
Description: Number of sugar-sweetened drinks consumed per day
Time Frame: Assessed as change between baseline well-child visit (WCV #1) and 24 month follow-up exit visit (well-child visit:WCV#3)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Number of Sugar Sweetened Beverages/Day
Arm/Group | CSM Theory-based Arm | AAP-based Arm
Number analyzed (Participants) | 357 | 365
Number of Sugar Sweetened Beverages/Day | 0.01 (0.88) | 0.04 (0.94)

5. Secondary Outcome: Change in Oral Health-related Quality of Life for Child
Description: Overall score on Early Childhood Oral Health Impact (ECOHIS) Scale with 13 items. Each item is on a Likert scale from 0 through 4. The overall score ranges from 0 to 52. An overall score was calculated for each child, and then a mean calculated for each arm of the study. Lower scores indicate a better oral health quality of life.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | CSM Theory-based Arm | AAP-based Arm
Number analyzed (Participants) | 357 | 380
scores on a scale | 0.56 (3.38) | 0.50 (3.42)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from baseline (WCV1) through the exit visit (WCV3).
Description: Adverse event information was collected for children, parent/caregivers and providers through communication with participants or family members when contact was made during study visits or during follow-up phone calls for data collection or retention purposes. Adverse events reported were unrelated to the study intervention. Adverse events were monitored after informed consent was received through study completion.
Groups:
- CSM Theory-based Arm Children: Children enrolled in the CSM theory-based didactic education and skills training Practice EMR changes arm
  CSM theory-based didactic education and skills training: Common-Sense Model of Self-Regulation (CSM) theory-based education and skills training for the provider to teach him/her to communicate core oral health facts to parents, provide a prescription to take their child to the dentist together with a list of Medicaid-accepting dentists in the area, and document the oral health encounter in EMR.
  Practice EMR changes: Enhancements to the EMR system to include oral health documentation (four questions) which will be implemented prior to enrolling any parent/caregiver and child participants into the study.
- CSM Theory-based Arm Parents/Caregivers: Parents/Caregivers enrolled in the CSM theory-based didactic education and skills training Practice EMR changes
  CSM theory-based didactic education and skills training: Common-Sense Model of Self-Regulation (CSM) theory-based education and skills training for the provider to teach him/her to communicate core oral health facts to parents, provide a prescription to take their child to the dentist together with a list of Medicaid-accepting dentists in the area, and document the oral health encounter in EMR.
  Practice EMR changes: Enhancements to the EMR system to include oral health documentation (four questions) which will be implemented prior to enrolling any parent/caregiver and child participants into the study.
- CSM Theory-based Arm Providers: Providers enrolled in the CSM theory-based didactic education and skills training Practice EMR changes
  CSM theory-based didactic education and skills training: Common-Sense Model of Self-Regulation (CSM) theory-based education and skills training for the provider to teach him/her to communicate core oral health facts to parents, provide a prescription to take their child to the dentist together with a list of Medicaid-accepting dentists in the area, and document the oral health encounter in EMR.
  Practice EMR changes: Enhancements to the EMR system to include oral health documentation (four questions) which will be implemented prior to enrolling any parent/caregiver and child participants into the study.
- AAP-based Arm Children: Children enrolled in the AAP-based didactic education
  AAP-based didactic education: American Academy of Pediatrics (AAP) based oral health education and follow the usual care for oral health assessment recommended by AAP guidelines.
- AAP-based Arm Parents/Caregivers: Parents/Caregivers enrolled in the AAP-based didactic education
  AAP-based didactic education: American Academy of Pediatrics (AAP) based oral health education and follow the usual care for oral health assessment recommended by AAP guidelines.
- AAP-based Arm Providers: Providers enrolled in the AAP-based didactic education
  AAP-based didactic education: American Academy of Pediatrics (AAP) based oral health education and follow the usual care for oral health assessment recommended by AAP guidelines.
Arm/Group | CSM Theory-based Arm Children | CSM Theory-based Arm Parents/Caregivers | CSM Theory-based Arm Providers | AAP-based Arm Children | AAP-based Arm Parents/Caregivers | AAP-based Arm Providers
All-Cause Mortality (participants affected / at risk) | 0/517 | 2/517 | 0/27 | 0/506 | 0/506 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/517 | 2/517 | 0/27 | 0/506 | 0/506 | 0/35
Other Adverse Events (participants affected / at risk) | 0/517 | 0/517 | 0/27 | 0/506 | 0/506 | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSM Theory-based Arm Children (N=517) | CSM Theory-based Arm Parents/Caregivers (N=517) | CSM Theory-based Arm Providers (N=27) | AAP-based Arm Children (N=506) | AAP-based Arm Parents/Caregivers (N=506) | AAP-based Arm Providers (N=35)
Death (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
As with any longitudinal studies there was follow-up losses at WCV2 and WCV3. But in the sample size calculation we accounted for 25% follow-up losses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/29/NCT03385629/Prot_SAP_000.pdf